CLINICAL TRIAL: NCT03364361
Title: Acupuncture for Perceived Stress in Military Personnel: A Feasibility Study
Brief Title: Acupuncture for Perceived Stress in Military Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Jane J. Abanes, Principal Investigator, United States Naval Medical Center, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NHCP. 2017.0057
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Acupuncture; Perceived Stress; Military Personnel
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acupuncture (Other): Feasibility Study
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Participants will receive a six-point standardized stress acupuncture (SSA) treatment once a week for 4 weeks. The SSA consists of GV- 20, GV-24.5 (Yin Tang), bilateral LI-4, and bilateral LR-3. This acupuncture protocol has been used as an effective treatment for stress-related symptoms in the operational theater.

SUMMARY:
Introduction: Although the physiologic response to stress is necessary for mammals to survive, prolonged stress response as a result of perceived stress can lead to allostatic load and loss of resilience to future stressors. To mitigate the consequences of allostatic load, researchers have investigated the effects of acupuncture as a promising intervention.

Objectives/Aims: The purpose of this study is to explore the feasibility and effect of a standardized stress acupuncture (SSA) approach on perceived stress in U.S. military personnel. Specific aims include the following: a) to determine feasibility of recruitment for SSA and implementation of study procedures in preparation for a methodologically rigorous study, b) to determine the acceptability of SSA treatment in a sample of military personnel with perceived stress, and c) to assess perceived stress and general health before and after SSA.

Methods and Analysis: This is a single-arm, single-site study protocol to assess feasibility of SSA in a total of 15 patients with perceived stress. Upon IRB approval and written informed consent, the participants will receive 4 weekly sessions of SSA which consists of 6 acupuncture points. Demographic information and attrition of participants will be monitored throughout the study. Patient-reported questionnaires including Acupuncture Expectancy Scale, Perceived Stress Scale, and SF-36 will be administered at baseline and then at the completion of the study. Descriptive statistics, reliable change indices (RCI), and Wilcoxon Signed-Ranks tests will be conducted to assess the magnitude of changes in scores.

Military Relevance: The three most common disability conditions in the military include musculoskeletal, psychiatric, and neurological body systems. Among these problems, however, mental health disorders remain a significant contributor to disability and suicide. Given the role of perceived stress in disability and suicidality in the military, intervening early before service members become at risk for severe injuries, hospitalizations, and chronic disability could help decrease burdensome problems.

DETAILED DESCRIPTION:
SPECIFIC OBJECTIVES:

Aim 1a: To determine feasibility of recruitment in service members for SSA. Expected Outcome: Participants will agree to receive SSA treatment for their perceived stress.

Aim 1b: To determine feasibility of implementation of study procedures including the following (Lancaster et al., 2004):

1. Inclusion and exclusion criteria.
2. Consent form procedures.
3. Storage and testing of equipment and materials (i.e., use of acupuncture needles, videotaping procedures, peer review feedback, randomization of peer review sessions, and use of a secure system for data management).
4. Training of staff in the administration of questionnaires and informed consent process.
5. Testing out the administration of data collection forms and questionnaires. Expected Outcome: The primary investigator (PI) will record field notes and report lessons learned in preparation for a trial with methodological rigor.

Aim 2: To determine the acceptability of SSA treatment in a sample of military personnel with perceived stress using the Acupuncture Expectancy Scale (AES) (Mao, Xie, & Bowman, 2010).

Expected Outcome: Participants will report SSA to be acceptable as a treatment for perceived stress.

Aim 3: To assess perceived stress and general health before and after SSA using the Perceived Stress Scale (PSS) (Cohen et al., 1983) and Short Form (SF) Health Survey-36 (Ware & Sherbourne, 1992) in the sample of patients who are receiving an SSA protocol.

Expected Outcome: Participants will report improved PSS and SF-36 scores at the completion of acupuncture treatment compared with baseline scores.

RESEARCH DESIGN:

1. General Approach:

   This is a single-arm, single-center pilot feasibility study in Naval Hospital Camp Pendleton's (NHCP) Branch Health Clinic (BHC) Yuma, Arizona. Service members who participate in this study will receive acupuncture for a total of four weeks. Because this is a feasibility study, there is no planned randomization or group comparison in this study. Convenience sampling will be used to recruit participants.
2. Description:

   Acupuncture is currently being performed as a treatment for musculoskeletal and psychological problems at BHC, Yuma.
3. Methods:

Procedures:

Research Team. The following personnel will comprise the research team for this study:

1. The PI is a licensed, credentialed PMHNP who is privileged to perform acupuncture at NHCP. The PI has performed acupuncture as an adjunct treatment for mental health problems including combat-related PTSD in active duty service members. The PI received her PMHNP education from universities in the U.S. and her acupuncture training and certification from Helm's Medical Institute's Medical Acupuncture for Physicians course.
2. The PhD-prepared licensed clinical psychologist received her doctorate degree from Uniformed Services University of Health Sciences. The psychologist is skilled to recruit and screen eligible participants, conduct informed consent, and provide questionnaires. She will be trained about the study's logistics and procedures.
3. The psychiatric technician received his education in the U.S. Navy. The technician is skilled to provide questionnaires and will be trained about the study's logistics and procedures.
4. The peer reviewer is an expert licensed, privileged acupuncturist at NHCP. She is a credentialed acupuncturist, has performed acupuncture for 4 years.

Training. Upon IRB approval, the research team will be trained on the following research activities: recruitment, screening of eligible participants, proper procedures when there are adverse events and psychological distress, informed consent process, follow-up tracking procedures, and administration of surveys and questionnaires.

The study staff (i.e., mentor and psychiatric technician) working with the PI will be required to undergo a special training prior to the beginning of the study to ensure consistency in study logistics and practices. The training will include logistics about the study such as participant check-in, study questionnaires, vital signs procedures, and follow-up periods. The PI will assess the study staff's research practices by enactment of skills and direct observation of these skills by the PI prior to study implementation. The PI will monitor all research activities conducted by the study staff throughout the study.

Eligibility Screening. Interested participants will be asked to call the mental health clinic to speak with the psychiatric technician, psychologist, or PI for screening. Screening of eligible participants will be conducted by the study staff via telephone or in-person at a private office in the mental health clinic at BHC, Yuma. Upon determination of eligibility, the participant will go through the informed consent process with the study staff in a private office located in the mental health department.

Baseline Survey. Participants will check-in in the mental health clinic where acupuncture treatments typically take place. Participants will fill out paper questionnaires upon check-in such as the demographic form, AES, PSS, and SF-36 survey prior to the initiation of the first acupuncture treatment.

Measures:

Participants will complete a demographics form and the following measures upon consent and enrollment in the study.

Demographics: Age; marital status; race; education level; and military characteristics (i.e., rank, branch of service, years of service, type of deployment, and times deployed) will be obtained at the beginning of the study using a self-report form.

Vital Signs (VS): Blood pressure (BP) of the right arm and heart rate measurements will be obtained before each treatment, about five minutes after the participant's arrival to the mental health clinic(Abdi et al., 2017). Vital signs will be measured by the research assistant using the vital signs mobile unit that is currently being used in the clinic.

Data Collection and Storage:

De-identified data will be coded independently by the coders (i.e., PI and mentor) using Microsoft Excel spreadsheets. These spreadsheets will be uploaded and shared between the coders via a DoD secure system called SAFE (AMRDEC, 2016) (see 'protection of patient privacy' section for details about the system). After discussion and consensus between the coders, a final spreadsheet will be created. This final spreadsheet will be uploaded and retrieved from SAFE and imputed from Excel into IBM SPSS Statistics software, which will be stored in the PI's password-protected personal laptop computer.

Treatment Procedures:

Participants will receive 4 weekly acupuncture sessions. No other follow-up session will be conducted after all treatments have been completed.

Treatment Location. The intervention will take place in a designated, private acupuncture/exam room in BHC, Yuma. The acupuncture room has a sink to wash and dry hands before and after treating each participant.

Treatment Supply. Standard acupuncture supply will be used.

Acupuncture Needles:

1. SEIRIN J-Type Sj.20x30 will be used for GV-20 and GV-24.5.
2. SEIRIN L-Type Lc.20x40 will be used for LI-4 and LR-3.

Treatment Protocol. Participants will receive a six-point SSA treatment once a week for 4 weeks. The SSA consists of GV- 20, GV-24.5 (Yin Tang), bilateral LI-4, and bilateral LR-3. This acupuncture protocol has been used as an effective treatment for stress-related symptoms in the operational theater (Koffman, 2011).

Statistical Analysis:

Sample Size Estimation. Given that this is a feasibility study, a sample size determination through statistical power calculations will not be conducted(Leon, Davis, & Kraemer, 2011). Obtaining a sample of 15 participants to complete the treatments will be the goal for this study. Fifteen is selected based on the short recruitment time frame (i.e., no more than two months) for this study. At least 20 will be recruited to account for potential missing data and attrition.

Missing Data. Randomly missing responses to items within the study's standardized measures (i.e., AES, PSS, SF-36) will be handled according to the scoring protocols of the measures. Details of any loss to follow-up will be evaluated to determine if they are based on study conditions, participant characteristics, or occupational demands. Because of the limited sample size, missing values will not be imputed.

Data Analysis. De-identified study data will be exported from Microsoft Excel into IBM SPSS Statistics software for analyses. Feasibility summaries and effect sizes will be the primary goals of the analyses; however, any tests of statistical significance will maintain an alpha of 0.05 (p < 0.05 for Type I error).

Aim 1a: Descriptive statistics will be used to describe the following: a) the sample, b) critical demographic, and service information of the participants, c) the number of individuals screened for the study versus the number of participants, and d) the number of participants who completed all visits versus the number of participants who withdrew from the study.

Aim 1b: The analysis of this aim will be qualitative in nature. At the end of the study, a text summary of feasibility of study procedures will be provided to delineate field notes and lessons learned in the implementation of this study.

Aim 2: Scores on the AES at baseline and then at the end of the study will be summarized using descriptive statistics. Change in the scores between the two times of assessment will also be generated and summarized. Wilcoxon Signed-Ranks tests will test the statistical significance of the change.

Aim 3: Descriptive statistical and graphical summaries of the PSS and SF-36 scores at baseline and end-of-study, as well as change in the scores between the two times of assessment will be evaluated. Given measurement error inherent in psychosocial measures, reliable change indices (RCI) will be generated for the PSS and each of the SF-36 measures. The RCI was originally proposed by Jacobson, Follette, and Revenstroff(Jacobson, Follette, & Revenstorf, 1984) and amended by Christensen and Mendoza(Christensen & Mendoza, 1986) as a measure of whether the change in an individual's score was significant (both statistically and clinically), after taking into account the reliability of the measure. An RCI value will be calculated for each participant for each coping and adjustment measure by subtracting the individual's baseline score from their respective post-intervention score then dividing by the standard error of the difference in the test. Calculation of the standard error of the difference for each measure used the direct method proposed by Jacobson and Traux(Jacobson & Truax, 1991). Published normative test-retest reliability coefficients for each of the standardized PSS and SF-36 measures in this study will be used in the calculation of the standard errors of the differences. The RCI values will then be summarized for reliable estimates of the effect of the acupuncture treatment on self-reported stress and general health. Wilcoxon Signed-Ranks tests will test the statistical significance of the change.

ELIGIBILITY:
Inclusion Criteria:

* Active duty service members will be considered eligible upon meeting the following criteria: 18 to 65 years of age, Self-report of perceived stress for at least one month. A score of 16 or above on the PSS. The choice of 16 on the PSS scale, as an eligibility criterion, was based on previous studies that use the same score criterion to describe the impact of perceived stress on allostatic load and the effect of acupuncture for perceived stress (Groer et al., 2016; Schroeder et al., 2017). Stable on psychiatric and other medications for at least three months. Able to sign an informed consent.

Exclusion Criteria:

* Recent medical surgery within one month; Alcohol abuse or dependence diagnosis within one month and active substance use/abuse/dependency treatment within one month; Pregnant women. Acupuncture can result in an induction of labor and spontaneous abortion in rare occasions(White et al., 2008); Has had acupuncture treatment in the past month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Descriptive statistics and Qualitative Text Summary | Throughout the study (4 weeks)
  Descriptive statistics will be used to describe the following: a) the sample, b) critical demographic, and service information of the participants, c) the number of individuals screened for the study versus the number of participants, and d) the number of participants who completed all visits versus the number of participants who withdrew from the study. The analysis of this aim will be qualitative in nature. At the end of the study, a text summary of feasibility of study procedures will be provided to delineate field notes and lessons learned in the implementation of this study.

SECONDARY OUTCOMES:
Acupuncture Expectancy Scale (AES) | Baseline and posttreatment measure at week 4.
  The AES is a 4-item questionnaire that measures the participants' expected responses to acupuncture. Participants' expected improvement from acupuncture is rated in a 5-point Likert-type scale ranging from not at all agree to completely agree (Mao et al., 2010). The total possible scores for AES range from 4 to 20, with higher scores indicating greater expectancy. In an initial validation, the instrument's Cronbach's alpha is .82 (Mao et al., 2007). The AES has been found to be reliable, valid, and has acceptable sensitivity to change during treatment starting at week 4 of treatment with increasing statistically significant changes with more acupuncture treatments (Mao et al., 2010).
Perceived Stress Scale (PSS) | Baseline and posttreatment measure at week 4.
  The PSS is a 10-item scale that has been used to evaluate perceived stress experience in adults (Cohen et al., 1983). Perceived general stress is rated in a 5-point Likert-type scale ranging from a never to very often. The total possible scores for PSS range from 0 to 56, with higher scores indicating higher stress. In a normative sample, the instrument's Cronbach's alpha is from .84 to .86 (Cohen et al., 1983).
Short Form-36 Health Survey | Baseline and posttreatment measure at week 4.
  The SF-36 is a 36-item scale that measures the multidimensional concept of health including perceptions about general health, physical health, mental health, and social functioning (Ware & Sherbourne, 1992). The questionnaire has been widely used in both clinical practice and research including in a sample of veterans (Kazis et al., 2004). The instrument has an internal consistency ranging from .52 to .89 (Kazis et al., 2004). This measure has moderate sensitivity in detecting changes in group scores using all SF-36 subscales (Busija, Osborne, Nilsdotter, Buchbinder, & Roos, 2008).

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center, San Diego, California, United States